CLINICAL TRIAL: NCT00309725
Title: Placebo-Controlled Evaluation of Galantamine in the Treatment of Alzheimer's Disease: A Cardiac Safety Study.
Brief Title: A Cardiac Safety Study of Galantamine in the Treatment of Alzheimer's Disease.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR012118
Record Dates: First submitted 2006-03-31; First posted 2006-04-03 (Estimated); Last update posted 2011-05-18 (Estimated); Status verified 2011-01

CONDITIONS: Alzheimer's Disease
Keywords: Alzheimer's Disease; cardiac arrhythmias
MeSH Terms: conditions — Alzheimer Disease; Arrhythmias, Cardiac | interventions — Galantamine

INTERVENTIONS:
Drug: galantamine

SUMMARY:
The objective of this trial was to investigate the effect of galantamine (an acetylcholinesterase inhibitor) on heart rate and PR interval (the time it takes for the heart's electrical impulse to get from the atria to the ventricles) during the administration of rapidly increasing doses and at the end of a 2-week treatment period with 32 mg per day in patients with Alzheimer's disease.

DETAILED DESCRIPTION:
This 6-week, double-blind, parallel group trial was also designed to detect cardiac arrhythmias and conduction disturbances, such as heart block. Holter monitors and Electrocardiograms were used to measure cardiac parameters at baseline, at the end of Week 2 (first dose of 12 mg twice daily), at the end of Week 4 (first dose of 16 mg twice daily) and at Week 6 (after 2 weeks of maximum tolerated dose allowed in the trial, i.e., 24 or 32 mg/day). Other safety data collected were adverse event reports, urine and blood analysis, vital signs and physical examination. Drug levels in the blood were also tested. Patients were randomized to receive either placebo or galantamine up to 32 mg daily (i.e., 4 mg twice daily in Week 1, 8 mg twice daily in Week 2, 12 mg twice daily in Weeks 3 and 4, and 16 mg twice daily in Weeks 5 and 6). Dosage could be reduced from 16 mg twice daily to 12 mg twice daily during the first 3 days of the 32 mg/day dosing period, if a patient could not tolerate the higher dose. This titration is more rapid and the dose is higher than currently recommended for treatment.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients diagnosed with Alzheimer's disease in accordance with NINCDS-ADRDA (National Institute of Neurological and Communicative Diseases and Stroke/Alzheimer's Disease and Related Disorders Association) classification for probable Alzheimer's disease
* Mild/moderate dementia as evidenced by a Mini-Mental State Examination (MMSE) score ranging from 11 to 24, inclusive, at baseline
* History of cognitive decline that has been gradual in onset and progressive over a period of at least 6 months
* Evidence of sustained memory deterioration in an otherwise alert patient, plus additional impairment in at least one of these five areas: orientation, judgment and problem-solving, functioning in community affairs, functioning in home and hobbies, and functioning in personal care
* Patients who live with or have regular daily visits from one or more responsible caregiver who are capable of assisting with the patient's medication, able to accompany the patient for assessments, and willing to provide information about the patient.On days that the patient was sent home with a Holter monitor, the caregiver was required to stay with the patient in the same household for the 24 hour duration of the cardiac assessment to ensure that the monitor lead placement remained intact. The caregiver was to be available the following day for the return of the Holter monitoring device
* Patient or patient's relative, guardian or legal representative have signed the informed consent.

Exclusion Criteria:

* Disorders such as Parkinson's disease, Pick's disease, or Huntington's chorea, Down's syndrome, Creutzfeldt-Jakob disease, Cushing's syndrome, or uncontrolled diabetes
* Cognitive impairment resulting from trauma, injury, or hypoxia
* Infection
* Mental retardation or dementia or clinically active cerebrovascular disease
* Current, clinically significant cardiovascular disease that would limit the patient's ability to complete a six-week trial.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 139 (Actual)
Dates: Study Completion 1999-10 (Actual)

PRIMARY OUTCOMES:
Hourly mean heart rates and PR intervals during each of the 24-hour Holter monitoring periods; Twenty-four hour mean, minimum and maximum heart rates and PR intervals during each of the 24-hour Holter monitoring periods

SECONDARY OUTCOMES:
Pharmacokinetics and other safety parameters including ECG parameters were other parameters of interest.

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- [Derived] Lim AWY, Schneider L, Loy C. Galantamine for dementia due to Alzheimer's disease and mild cognitive impairment. Cochrane Database Syst Rev. 2024 Nov 5;11(11):CD001747. doi: 10.1002/14651858.CD001747.pub4. PMID 39498781
- See also: A Cardiac Safety Study of Galantamine in the Treatment of Alzheimer's Disease — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=742&filename=CR012118_CSR.pdf